CLINICAL TRIAL: NCT05794984
Title: Targeted Focus Groups Discussions (FGDs) and Cross-sectional Questionnaire to Address Questions Regarding Telemedicine Concept and Knowledge, and Social Media Usage Among People Who Inject Drugs (PWID) in Greece
Brief Title: Telemedicine and Social Media for People Who Inject Drugs (PWID) in Greece
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Hellenic Scientific Society for the Study of AIDS, Sexually Transmitted and Emerging Diseases (Other)
Responsible Party: Principal Investigator, Andrew Talal, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00007088
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Drug Abuse, Intravenous; Internet; Social Media; Telemedicine
MeSH Terms: conditions — Substance Abuse, Intravenous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Targeted Focus Group Discussions and Cross-sectional questionnaire: 57 people for targeted Focus Group Discussions 162 people for Cross-sectional questionnaire
  Interventions: Other: Focus group discussions and survey questionnaire

INTERVENTIONS:
Other: Focus group discussions and survey questionnaire — Questions regarding internet and social media usage, as well as telemedicine concept and knowledge. Assessment of the feasibility, acceptability and accessibility of social media and telemedicine as methods to obtain healthcare. Perceptions for high-quality healthcare access, confidentiality, privacy, and security, will also be explored.

SUMMARY:
The current study seeks to address questions regarding internet and social media usage as well as telemedicine concept and knowledge, by conducting targeted focus group discussions (FGDs) and administering cross-sectional questionnaires among PWID in Greece. Further parameters, such as perceptions for high-quality healthcare access, confidentiality, privacy, and security, will also be explored.

DETAILED DESCRIPTION:
The study's aim is to access the feasibility, acceptability and accessibility of social media and telemedicine as methods to obtain healthcare, in order to improve linkage-to-care among Greek substance users. Underserved populations, such as people who inject drugs (PWID) have limited access to healthcare and a potential solution to expanding healthcare access points is telemedicine. For the past decade, the investigators have studied the efficacy of a facilitated telemedicine model for hepatitis C virus (HCV) treatment integrated into opioid treatment programs (OTPs) for PWIDs. The investigators have achieved high rates of HCV resolution and high patient-satisfaction through facilitated telemedicine. The investigators now seek to explore whether this same intervention might be feasible and acceptable in Greece. The first step is to capture and explore the current knowledge, experiences, believes, perceptions and attitudes of PWID in Greece regarding internet and social media usage and telemedicine concept, through targeted Focus Group Discussions (FGDs) and administration of cross-sectional questionnaire. The perceptions for high-quality healthcare, confidentiality, privacy and security matters will also be explored as well as further relevant attributes.

ELIGIBILITY:
Inclusion Criteria for the FDGs:

* >18 years old
* PWID
* Willing and able to provide informed consent and participate
* Fluent in Greek spoken language
* Internet access

Inclusion Criteria for the cross-sectional questionnaire:

* >18 years old
* PWID
* Willing and able to provide informed consent and participate
* Fluent in Greek spoken language

Exclusion Criteria for FGD and cross-sectional questionnaire:

* <18 years old
* Unable/unwilling to consent
* Legally incompetent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PWID are a medically and socially vulnerable population with high incidence of overdose, mental illness and infections such as HIV and hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
There are not specific predetermined endpoints to be defined. | For the FGDs approximately up to 3-4 months is needed to enroll all study subjects. For the cross-sectional questionnaire approximately up to 6-8 months is needed to enroll all study subjects. Endpoints will be generated according to study's results.
  This is a mixed methods study designed to assess the feasibility, acceptability, and accessibility of telemedicine and social media to improve healthcare access among Greek PWUD. It is not an interventional trial. The results of this study will be used to generate endpoints and sample sizes for a larger trial.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Talal, MD, Principal Investigator — University at Buffalo
Locations (1):
- Prometheus, Athens, Greece

REFERENCES:
- [Background] Talal AH, Andrews P, Mcleod A, Chen Y, Sylvester C, Markatou M, Brown LS. Integrated, Co-located, Telemedicine-based Treatment Approaches for Hepatitis C Virus Management in Opioid Use Disorder Patients on Methadone. Clin Infect Dis. 2019 Jul 2;69(2):323-331. doi: 10.1093/cid/ciy899. PMID 30329042
- [Background] Talal AH, McLeod A, Andrews P, Nieves-McGrath H, Chen Y, Reynolds A, Sylvester C, Dickerson SS, Markatou M, Brown LS. Patient Reaction to Telemedicine for Clinical Management of Hepatitis C Virus Integrated into an Opioid Treatment Program. Telemed J E Health. 2019 Sep;25(9):791-801. doi: 10.1089/tmj.2018.0161. Epub 2018 Oct 16. PMID 30325701
- [Background] Talal AH, Markatou M, Sofikitou EM, Brown LS, Perumalswami P, Dinani A, Tobin JN. Patient-centered HCV care via telemedicine for individuals on medication for opioid use disorder: Telemedicine for Evaluation, Adherence and Medication for Hepatitis C (TEAM-C). Contemp Clin Trials. 2022 Jan;112:106632. doi: 10.1016/j.cct.2021.106632. Epub 2021 Nov 20. PMID 34813962
- [Background] Talal AH, Sofikitou EM, Wang K, Dickerson S, Jaanimagi U, Markatou M. High Satisfaction with Patient-Centered Telemedicine for Hepatitis C Virus Delivered to Substance Users: A Mixed-Methods Study. Telemed J E Health. 2023 Mar;29(3):395-407. doi: 10.1089/tmj.2022.0189. Epub 2022 Aug 4. PMID 35925809
- [Background] Hatzakis A, Sypsa V, Paraskevis D, Nikolopoulos G, Tsiara C, Micha K, Panopoulos A, Malliori M, Psichogiou M, Pharris A, Wiessing L, van de Laar M, Donoghoe M, Heckathorn DD, Friedman SR, Des Jarlais DC. Design and baseline findings of a large-scale rapid response to an HIV outbreak in people who inject drugs in Athens, Greece: the ARISTOTLE programme. Addiction. 2015 Sep;110(9):1453-67. doi: 10.1111/add.12999. Epub 2015 Jul 14. PMID 26032121
- [Background] Sypsa V, Psichogiou M, Paraskevis D, Nikolopoulos G, Tsiara C, Paraskeva D, Micha K, Malliori M, Pharris A, Wiessing L, Donoghoe M, Friedman S, Jarlais DD, Daikos G, Hatzakis A. Rapid Decline in HIV Incidence Among Persons Who Inject Drugs During a Fast-Track Combination Prevention Program After an HIV Outbreak in Athens. J Infect Dis. 2017 May 15;215(10):1496-1505. doi: 10.1093/infdis/jix100. PMID 28407106
- [Derived] Papalamprakopoulou Z, Roussos S, Ntagianta E, Triantafyllou V, Kalamitsis G, Dharia A, Sypsa V, Hatzakis A, Talal AH. Considerations for equitable distribution of digital healthcare for people who use drugs. BMC Health Serv Res. 2025 Apr 10;25(1):531. doi: 10.1186/s12913-025-12619-7. PMID 40211324
- [Derived] Papalamprakopoulou Z, Ntagianta E, Triantafyllou V, Kalamitsis G, Dharia A, Dickerson SS, Hatzakis A, Talal AH. Telehealth to increase healthcare access; perspectives of people who use drugs. BMC Med Inform Decis Mak. 2024 Oct 19;24(1):306. doi: 10.1186/s12911-024-02718-6. PMID 39425182
- See also: Extensions of Respondent-Driven Sampling: Analyzing Continuous Variables and Controlling for Differential Recruitment — http://www.respondentdrivensampling.org/reports/steering.pdf